CLINICAL TRIAL: NCT01487824
Title: What is the Impact of Early Life Exposures on the Cardiovascular System in Young Adulthood? A 25-Year Follow-up Study of Preterm-born Individuals
Brief Title: What is the Impact of Early Life Exposures on the Cardiovascular System in Young Adulthood?
Acronym: EVS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: Early Vascular Study
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2012-06

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, immortalised cell lines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm-born Young Adults
- Term-born Young Adults

SUMMARY:
The purpose of this study is to investigate whether early life exposures such as premature birth or exposure to preeclampsia before you are born results in long-term alterations in the cardiovascular system that increase risk of cardiovascular disease development.

DETAILED DESCRIPTION:
While the incidence of cardiovascular disease has reduced dramatically, coinciding with favourable changes in risk factors, cardiovascular disease remains the single largest cause of mortality and premature mortality in the United Kingdom. Identification of novel biological pathways that underlie disease susceptibility raises the potential for new early primary prevention strategies to complement classical management. There is particular interest in the role of early environment in 'programming' risk of cardiovascular disease in later life and growing evidence that various early life exposures impact cardiovascular health in the longer term.

We have thus designed the Early Vascular Study to investigate the long-term impact of early life exposures, with a particular focus on the impact of preterm birth, in the presence or absence of pregnancy-induced hypertension in the mother, on the cardiovascular system in young adulthood. This study also allows investigation of the long term impact of perinatal interventions used in this cohort. Comprehensive multi-modality non-invasive imaging measures of cardiovascular structure and function allow precise quantification of cardiovascular phenotype. This is combined with blood sample collection to study changes in molecular and metabolic markers and pathways.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Preterm-born Cohort: Born premature (<37 weeks completed gestation), originally recruited as part of a randomised feeding trial at birth from one of five United Kingdom centres between 1982 and 1985.
* Term-born Cohort: Born at term (>37 weeks completed gestation) with normal birth weight for gestational age.
* Able (in the Investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

-The participant may not enter the study if ANY of the following apply:

* Unwilling or unable to give informed consent for participation in the study.
* Any significant disease or disorder which, in the opinion of the investigator, might influence the participant's ability to participate in the study.
* Contraindication to Cardiovascular Magnetic Resonance Imaging.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Preterm-born Cohort: A cohort of preterm-born young adults who were enrolled, at birth, from five centres in England between 1982 and 1985 into a randomised trial of milk feeding regimes to study the influence of early diet on later cognitive function and cardiovascular disease.
  Term-born Cohort: A cohort of controls born at term with normal birthweight now aged between 20 and 40 years to provide age stratified normal ranges for the outcome measures.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cardiac structure | Young adulthood
  Left ventricular mass

SECONDARY OUTCOMES:
Cardiac function | Young adulthood
  Global longitudinal strain and diastolic strain rate
Arterial stiffness | Young adulthood
  Pulse wave velocity
Microvascular structure | Young adulthood
  Capillary density
Cardiac structure | Young Adulthood
  Right ventricular mass

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, PhD, MRCP, Principal Investigator — Oxford Cardiovascular Clinical Research Facility, Department of Cardiovascular Medicine, University of Oxford
Locations (1):
- Cardiovascular Clinical Research Facility, Dept of Cardiovascular Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Lewandowski AJ, Lamata P, Francis JM, Piechnik SK, Ferreira VM, Boardman H, Neubauer S, Singhal A, Leeson P, Lucas A. Breast Milk Consumption in Preterm Neonates and Cardiac Shape in Adulthood. Pediatrics. 2016 Jul;138(1):e20160050. doi: 10.1542/peds.2016-0050. Epub 2016 Jun 14. PMID 27302980
- [Derived] Lewandowski AJ, Augustine D, Lamata P, Davis EF, Lazdam M, Francis J, McCormick K, Wilkinson AR, Singhal A, Lucas A, Smith NP, Neubauer S, Leeson P. Preterm heart in adult life: cardiovascular magnetic resonance reveals distinct differences in left ventricular mass, geometry, and function. Circulation. 2013 Jan 15;127(2):197-206. doi: 10.1161/CIRCULATIONAHA.112.126920. Epub 2012 Dec 5. PMID 23224059